CLINICAL TRIAL: NCT01792791
Title: Assessment of Biomarkers Associated With Joint Injury and Subsequent Post-Traumatic Arthritis
Brief Title: Post-traumatic Arthritis Associated With Joint Injury
Status: Completed | Type: Observational
Sponsor: Duke University (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: Pro00038254
Record Dates: First submitted 2012-10-25; First posted 2013-02-15 (Estimated); Last update posted 2016-12-19 (Estimated); Status verified 2015-08

CONDITIONS: Arthritis
MeSH Terms: conditions — Arthritis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Single Arm
  Interventions: Procedure: Tissue sample collection at the time of surgery

INTERVENTIONS:
Procedure: Tissue sample collection at the time of surgery — Spanning surgery
  * A blood sample (32.5 ml)
  * joint aspirate (removal of synovial fluid) from both knees
  * urine sample
  ORIF surgery
  * Joint aspirate (removal of synovial fluid) from both knees
  * A blood sample (32.5 ml)
  * Urine Sample
  If patients only require one surgery, sample will be collected only once.

SUMMARY:
Arthritis is the nation's most common cause of disability. An estimated 50 million U.S. adults (about 1 in 5) report doctor-diagnosed arthritis. Twenty three million U.S. adults of working age (18-64 years) have arthritis; and in this age group arthritis-attributable work limitations affect about 1 in 3 people. An estimated 12% of all patients seeking intervention for symptomatic arthritis have an etiology of previous trauma to the involved joint.

The purpose of this study is to examine these inflammatory compounds in the joint fluid (synovial fluid), the joint lining (synovium), and in blood among subjects with isolated intra-articular fractures.

The hypothesis is that early levels of intra-articular inflammation and markers of joint tissue degeneration following articular fracture in the human knee are predictive of the development of PTA (Post Traumatic Arthritis). Early levels of intra-articular inflammation and markers of joint tissue degeneration identified from human knee joints following articular injury are predictive of the development of PTA in the mouse knee.

Samples of blood, urine and synovial fluid will be taken at the spanning frame surgery and only synovial fluid at the ORIF (Open Reduction Internal Fixation)surgery. Two MRIs (Magnetic Resonance Imaging) will be part of this study at 4 weeks and 18 months.Participants will complete a set of questionnaires(KOOS: Knee Injury and Osteoarthritis Outcome Score) at 4 weeks and 18 months.

DETAILED DESCRIPTION:
40 patients with a closed unilateral articular fracture of the knee requiring operative treatment will be enrolled over an 18 month period. Tissue samples including synovial fluid from the injured and contralateral knee, serum and urine will be collected pre-operatively at the time of framing and ORIF. If patients only need to have one surgery (ORIF) sample will be collected only once. MRI imaging of the injured knee will be obtained after fixation at between week 6 and 8 and at 18 months. Tissue samples will be analyzed for established biomarkers of joint inflammation and degradation. Patients will be followed for 18 months to assess for signs of post-traumatic arthritis. Imaging with plain film and MRI will occur at 18 months. MRI imaging analysis of cartilage thickness and composition changes will be assessed in the injured knees. Assessment of articular cartilage and joint space narrowing and KOOS will be correlated to biomarkers that may be indicative and predictive of joint degeneration and the development of PTA.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be adult patients (over 18 years old)
* Patients must present with a unilateral closed intra-articular fracture of the knee.

Exclusion Criteria:

* Pre-existing arthritis in the injured or contra-lateral knee,
* Previous total knee replacement
* Active joint infection
* Pathologic fracture
* Active inflammatory arthritis
* Open fracture of the involved knee
* Contra-lateral knee injury
* HIV infection (if previously known)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults that are at least 18 years old and had a unilateral closed intra articular fracture of the knee that requires surgery.
Sampling Method: Probability Sample
Enrollment: 20 (Actual)
Dates: Start 2012-10; Primary Completion 2016-11 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Markers of joint tissue degeneration following articular fracture | 18 months after Injury
  Tissue samples will be collected at the time of surgery and they will be taken to Duke Basic Science lab where they will be analyzed.

SECONDARY OUTCOMES:
KOOS questionnaire | Participants will complete this questionnaire at the 18 month follow up
  Participants will be scheduled for an MRI 18 months after surgery and a questionnaire will be completed at that time.

OTHER OUTCOMES:
Change from baseline at 18 months of the extracellular matrix and morphology of knee cartilage using MRI | Between week 2 and 6 and at 18 months after definitive fixation
  Two MRIs will be scheduled for all the study participants at 4 weeks (with a 2-6 weeks window) and at 18 months.

CONTACTS AND LOCATIONS:
Overall Officials: Steven Olson, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States